CLINICAL TRIAL: NCT00703417
Title: Does Bone Structure Explain the Increased Fracture Risk in Type II Diabetes Patients? A Pilot Study
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Thomas M. Link, M.D., University of California, San Francisco
Other Study IDs: Diabetes
Record Dates: First submitted 2008-06-19; First posted 2008-06-23 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2011-06

CONDITIONS: Osteoporosis
Keywords: osteoporosis; diabetes
MeSH Terms: conditions — Osteoporosis; Diabetes Mellitus | interventions — Magnetic Resonance Imaging; Tomography, X-Ray Computed

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: Healthy post-menopausal women
  Interventions: Device: magnetic Resonance Imaging; Device: High resolution peripheral quantitative computed tomography
- 2: Diabetic without fracture
  Interventions: Device: magnetic Resonance Imaging; Device: Computed Tomography; Device: High resolution peripheral quantitative computed tomography
- 3: Diabetic with fracture
  Interventions: Device: magnetic Resonance Imaging; Device: Computed Tomography; Device: High resolution peripheral quantitative computed tomography

INTERVENTIONS:
Device: magnetic Resonance Imaging — MRI of the calcaneus, the distal tibia, the distal radius and also lower back.
Device: Computed Tomography — CT scan of the lower back and hip
  Groups: 2; 3
Device: High resolution peripheral quantitative computed tomography — HR-pQCT of the distal radius and distal tibia

SUMMARY:
For this cross-sectional case control pilot study 30 women, 55-75 years old with type II diabetes will be recruited. Diabetes will be defined as self-report of diabetes previously diagnosed by a physician, use of hypoglycemic medications, or fasting glucose > 126 mg/dl (7.0mM) in accordance with the American Diabetes Association criteria. The diabetic patient population will be divided into 2 groups: patients with status post low energy fractures of the proximal humerus, the proximal femur, the ankle and the foot (n=10) versus diabetic patients with no fractures or low energy trauma fracture history (n=10). An additional group of 10 diabetic postmenopausal women will be recruited and will have magnetic resonance imaging (MRI) of the lower back only. Caucasian, Asian and Hispanic women will be combined since a previous study suggested that BMD is very similar in these 3 population and that ethnic differences are minimal. In addition a population of 10 age-matched, BMI-matched, race-matched healthy women, without osteoporotic fractures will be examined. In all of these volunteers a medical history will be obtained to ensure good health status and rule out chronic diseases that would have an impact on bone metabolism. Patients will undergo MRI, QCT and high-resolution peripheral quantitative computed tomography (HR-pQCT) examinations to determine bone mineral density and bone structure/quality.

The hypothesis of this pilot project is that type II diabetic patients with and without low-energy fractures have a different trabecular bone architecture and composition, which is also different when compared to normal age-matched healthy patients. Architectural differences in these three patient groups may be visualized with high resolution MRI and high-resolution peripheral quantitative computed tomography (HR-pQCT) and will be most pronounced at the calcaneus and the distal tibia. Analyzing structure parameters obtained from high resolution MRI and spectroscopy may improve our understanding of the pathophysiology of diabetic bone disease and the prediction of fracture risk in an elderly diabetic population.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal female, 55-75 years old
* History of Type II diabetes, as defined by the American Diabetes Association for more than 5 years that is either insulin requiring or treated with oral therapies such as sulfonylureas and metformin
* Body mass index (BMI) of 19-35
* Able to move without walkers and without a history of long periods (>3 months) of inactivity
* Additional Inclusion criteria for fracture participants:
* Fractures of the proximal humerus and femur as well as the ankle and foot should have occurred after the onset of diabetes and should have been caused by a low energy trauma such as falling from standing height. All fractures will be verified by radiographs.

Exclusion Criteria:

* Severe neuropathic disease such as neurogenic osteoarthropathies (i.e., Charcot joints) of the foot
* Steroid users or have disease conditions that could play a significant role in the development of osteoporosis such as idiopathic osteoporosis, immobilization, hyperparathyroidism, or hyperthyroidism
* Diseases that may affect bone metabolism: alcoholism, chronic drug use, chronic gastrointestinal disease, renal or hepatic impairment
* Chronic treatment with antacids, estrogen, adrenal or anabolic steroids, anticonvulsants, anticoagulants, or pharmacologic doses of Vitamin A supplements 6 months prior
* Diabetic patients on rosiglitazone or pioglitazone medications
* high energy trauma, e.g., due to motor vehicle accidents
* Pathological fractures of other origin, i.e., tumor, tumor-like lesions as well as focal demineralization visualized on radiographs
* History of fluoride, bisphosphonate, calcitonin or tamoxifen use
* History of unstable cardiovascular disease or uncontrolled hypertension
* MRI contraindications
* Body mass index greater than 35

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10 healthy postmenopausal women 10 postmenopausal women with Type II Diabetes and without fracture 10 postmenopausal women with Type II Diabetes and with fracture of the long bone of the upper arm, hip, ankle, or foot 10 postmenopausal women with Type II Diabetes with and without fracture
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2006-05; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- China Basin Imaging Center, San Francisco, California, United States